CLINICAL TRIAL: NCT02466100
Title: Goals of Care Communication in Advanced Heart Failure
Brief Title: Goals of Care Communication
Acronym: GoC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Cynthia M. Dougherty, Professor, Biobehavioral Nursing and Health Systems, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 44610-ED
Record Dates: First submitted 2014-11-07; First posted 2015-06-09 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Patient Care Planning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Goc Intervention (Experimental): Patient education materials, study nurse phone call, tip sheet, provider tip sheet
  Interventions: Behavioral: goals of care
- usual care (No Intervention): care as usual in the community

INTERVENTIONS:
Behavioral: goals of care — . Patients in the GoC intervention group, telephone coaching by a research nurse to help patients role-play talking with their HF providers. Both patients and their providers, will be provided with summaries of individualized, patient-centered information about patient preferences for communicating about end-of-life care and patient self-identified barriers to and facilitators of communication about end-of-life care with tips on how to initiate goals of care discussions. Providers of patients in the intervention group will also be provided with patient-specific prognostic information based on the Seattle Heart Failure Model.
  Arms: Goc Intervention

SUMMARY:
This study proposes to evaluate, among adults with advanced heart failure (HF) and their health care providers, the effects of a communication intervention designed to improve patient-provider communication about goals of care (GoC). Patient activated GoC conversations can result in providers' better understanding their patients' preferences for end-of-life care. GoC conversations that occur over time may allow patients and providers to consider a wider range of options earlier in the HF illness trajectory. Preliminary data suggests that the proposed GoC intervention increases the occurrence and quality of patient-provider communication about end-of-life care for advanced COPD. The proposed study will test the effects of the GoC intervention compared to usual care, using a randomized, 2-group (N = 80, n = 40/arm), repeated-measures design. Measures will be taken at a patient's baseline study entry and after the next scheduled clinic visit. Specific Aim 1 is to evaluate change in number of GoC conversations between patient and provider between the two groups. Specific Aim 2 is to examine whether the intervention increases patient quality of life, referrals to palliative care, advance care planning, decreases depression and anxiety. Specific Aim 3 is to describe the feasibility, acceptability, perceived benefits, burden, and implementation success of the intervention in the heart failure clinic setting. Patients will be randomized to the GoC intervention or to receive usual care. Patients in the GoC intervention group, telephone coaching by a research nurse to help patients role-play talking with their HF providers. Both patients and their providers, will be provided with summaries of individualized, patient-centered information about patient preferences for communicating about end-of-life care and patient self-identified barriers to and facilitators of communication about end-of-life care with tips on how to initiate goals of care discussions. Providers of patients in the intervention group will also be provided with patient-specific prognostic information based on the Seattle Heart Failure Model. The GoC intervention will be tested in a real-world clinic setting. This intervention is expected to be relatively cost-effective and easily translated into general cardiology practice in the future. The study is expected to make significant contributions to provision of earlier access to palliative care in the advanced HF disease trajectory.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of HF from either systolic or diastolic dysfunction, with an ejection fraction of ≤ 40%
2. Completion of an outpatient HF visit within the past 6 months
3. Ability to read, write, and speak in English

Exclusion criteria:

1. Short BLESSED cognitive score > 10 to rule out significant cognitive impairment;82
2. Diagnosis of any additional terminal illness with life expectancy of ≤ 1 year not related to heart disease
3. Psychiatric illness that required hospitalization in the past year; and (4) age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-06; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
quality of communication | 1 month after intervention completed
  qoc questionnaire

SECONDARY OUTCOMES:
HF qol | 1 month after intervention completed
  KCCQ questionnaire
anxiety | 1 month after intervention completed
  GAD-7 questionnaire
depression | 1 month after intervention completed
  phq-9 questionnaire
advanced directives | 1 month after intervention completed
  completion of adv directive or 5 wishes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Doorenbos AZ, Levy WC, Curtis JR, Dougherty CM. An Intervention to Enhance Goals-of-Care Communication Between Heart Failure Patients and Heart Failure Providers. J Pain Symptom Manage. 2016 Sep;52(3):353-60. doi: 10.1016/j.jpainsymman.2016.03.018. Epub 2016 Jul 9. PMID 27401505